CLINICAL TRIAL: NCT06040762
Title: The "Get Moving Trial": A Phase I/II RCT of Home-Based (P)Rehabilitation With ExerciseRx in Bladder Cancer and Upper Tract Urothelial Cancer
Brief Title: A Home-Based Prehabilitation Exercise Intervention for Improving Physical Function in Patients With Bladder Cancer and Upper Tract Urothelial Cancer, Get Moving Trial
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: Bladder Cancer Advocacy Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RG1123479; NCI-2023-05596 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); RG1123479 (Other: Fred Hutch/University of Washington Cancer Consortium); FHIRB0020171 (Other: Fred Hutch/University of Washington Cancer Consortium)
Record Dates: First submitted 2023-08-21; First posted 2023-09-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Bladder Cancer; Urothelial Carcinoma; Upper Tract Urothelial Carcinoma; Renal Pelvis and Ureter Urothelial Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms; Carcinoma, Transitional Cell | interventions — Practice Guidelines as Topic; Standard of Care; Interviews as Topic; Exercise Test

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A ([P]REHAB intervention) (Experimental): Starting at least 4 weeks prior to date of surgery, patients use the ExerciseRx app to follow the (P)REHAB exercise program, which consists of four 20-30 minute home exercise sessions per week and personalized step count goal setting and tracking, while receiving SOC chemotherapy, if applicable, prior to SOC surgery and for 90 days following surgery (total ~4-7 months). Patients also download the FitBit app and wear a FitBit throughout the study.
  Interventions: Other: Exercise Intervention; Other: App-Based Intervention; Other: Interview; Other: Wearable Activity Tracker; Other: Physical Performance Testing; Other: Questionnaire Administration
- Arm B (standard of care) (Active Comparator): Patients receive SOC educational materials and, starting at least 4 weeks prior to date of surgery, patients wear a FitBit and use the FitBit app while receiving SOC chemotherapy, if applicable, prior to SOC surgery.
  Interventions: Other: Best Practice; Other: App-Based Intervention; Other: Wearable Activity Tracker; Other: Physical Performance Testing; Other: Questionnaire Administration

INTERVENTIONS:
Other: Best Practice — Receive SOC educational materials
  Other Names: standard of care; standard therapy
  Arms: Arm B (standard of care)
Other: Exercise Intervention — Receive (P)REHAB exercise program
  Arms: Arm A ([P]REHAB intervention)
Other: App-Based Intervention — Use ExerciseRx app
  Arms: Arm A ([P]REHAB intervention)
Other: App-Based Intervention — Use FitBit app
Other: Interview — Ancillary studies
  Arms: Arm A ([P]REHAB intervention)
Other: Wearable Activity Tracker — Wear FitBit
Other: Physical Performance Testing — Ancillary studies
  Other Names: Physical Fitness Testing; Physical Function Testing
Other: Questionnaire Administration — Ancillary studies

SUMMARY:
Prehabilitation refers to the process of improving a patient's functional capabilities prior to a surgical procedure with the goal of decreasing post-surgical inactivity and physical decline. This clinical trial evaluates the utility of a personalized home-based prehabilitation exercise intervention for the improvement of physical function and surgical outcomes in patients with urothelial carcinoma undergoing definitive or consolidative surgery of the bladder (radical cystectomy) or upper tract (nephroureterectomy, ureterectomy) with or without preceding neoadjuvant/systemic therapy. The exercise intervention includes at-home exercise sessions focused on the improvement of core strength and balance as well as personalized step count goals, delivered to patients remotely via a smart-device-based application (ExerciseRx). Encouraging physical activity before surgery may improve physical function and surgical outcomes in patients who are scheduled to undergo surgery for their bladder or urothelial cancer.

DETAILED DESCRIPTION:
OUTLINE: Patients are randomized to 1 of 2 arms and are followed from enrollment through surgery, and for 90 days following surgery (total estimated time on study: ~4-7 months).

ARM A: Starting at least 4 weeks prior to date of surgery, patients use the ExerciseRx application (app) to follow the (P)REHAB exercise program, which consists of four 20-30 minute home exercise sessions per week approximately 4-6 weeks prior to surgery and personalized step count goal setting and tracking, while receiving standard of care (SOC) chemotherapy, if applicable, prior to SOC surgery, and for 90 days following surgery. Patients also wear a FitBit and use the FitBit app on study.

ARM B: Patients receive SOC educational materials and, starting at least 4 weeks prior to date of surgery, patients wear a FitBit and use the FitBit app while receiving SOC chemotherapy, if applicable, prior to SOC surgery.

After completion of study intervention, patients are followed up at 90 days following SOC surgery.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* English-speaking
* Planned treatment with radical cystectomy or radical nephroureterectomy/ureterectomy with or without preceding systemic therapy as indicated by the patient's surgeon with enough time to complete a minimum of 4 weeks of exercises before surgery if enrolled in the (P)REHAB arm
* Willing and able to participate in trial activities

Exclusion Criteria:

* Cognitive/mental impairment that will preclude ability to participate in routine exercise activities. Significant cognitive or memory impairment or baseline dementia that would preclude a patient's ability to follow instructions or reproduce exercises
* Immobility, inability/unwillingness to perform personalized exercise program. Inability to perform exercises safely from seated or standing position at home or recent falls or high fall risk. Neurologic or orthopedic condition(s) that restricts participation in unsupervised home exercises, such as prior stroke with neurologic impairment, weight-bearing precautions, or unwillingness to participate in exercises
* Participants who have nonmuscle-invasive urothelial cancer of the bladder/upper tract anticipating undergoing organ-preserving treatments, or radiographic evidence of metastatic disease involving other organs including brain metastases.
* Patients with predominant histology other than urothelial carcinoma of the bladder or upper tracts (e.g. metastasis from another cancer) who would not otherwise be considered candidates for standard definitive or consolidative surgeries (radical cystectomy, ureterectomy, radical nephroureterectomy) with/without treatment with preoperative/neoadjuvant systemic therapy.
* Uncontrolled or concurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study
* Inability to understand or read English
* Lack of access or lack of sufficient facility to use an Android or iOS smart device with the minimum criteria for using ExerciseRx
* Not receiving surgery at UWMC
* Participation in a clinical trial that does not permit enrollment in the Get Moving trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Trial recruitment | At enrollment
  Trial recruitment (proportion enrolled versus eligible, reason for not enrolling) will be described via qualitative report.
Trial retention | Through study completion, on average 4-7 months
  Trial retention (proportion retained versus all enrolled, reason for not completing) will be described via qualitative report. Successful retention is defined as continued participation within the trial until 4-7 months post enrollment (90 days post surgery) (T3).
Change in physical function | From enrollment (T1) to 1-4 months post enrollment (before surgery) (T2)
  Physical function will be measured by the Short Performance Physical Battery (SPPB). Change in physical function will be measured and compared between the (P)REHAB and standard of care arms. SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, potential cachexia, and mobility disability are determined to be disabled.
Change in physical function | From 1-4 months post enrollment (before surgery) (T2) to 4-7 months post enrollment (90 days post surgery) (T3)
  Physical function will be measured by the Short Performance Physical Battery (SPPB). Change in physical function will be measured and compared between the (P)REHAB and standard of care arms. SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, potential cachexia, and mobility disability are determined to be disabled.
Change in physical function | From enrollment (T1) to 4-7 months post enrollment (90 days post surgery) (T3)
  Physical function will be measured by the Short Performance Physical Battery (SPPB). Change in physical function will be measured and compared between the (P)REHAB and standard of care arms. SPPB scores range from zero to 12 possible points. SPPB score of 3-9 points in persons with possible sarcopenia but no mobility disability indicates frailty; SPPB score of 10 or greater for persons with no sarcopenia and no mobility disability indicates robustness. Persons with a score of 2 or lower who have sarcopenia, potential cachexia, and mobility disability are determined to be disabled.

SECONDARY OUTCOMES:
Protocol adherence | Through study completion, on average 7 months
  Protocol adherence (proportion adhered versus all enrolled, specifics for how protocol was not followed and why) will be described via qualitative report. Protocol adherence for the (P)REHAB arm is defined as completion of >=70% of all exercise activities (goal 4x weekly, 20-30min/session) as measured using the ExerciseRx app.
Patient experience with use of ExerciseRx app, including app engagement ([P]REHAB arm only) (feasibility) | Through study completion, on average 7 months
  Qualitative experience will be assessed by Zoom interviews (usability interview) with a subset of volunteer participants from the (P)REHAB arm and app engagement will be assessed by an affinity analysis of the MAUQ
Frailty | From enrollment (T1) to 3-4 months post enrollment (before surgery) (T2)
  Frailty will be assessed using the Cancer and Aging Resilience Geriatric Assessment.
Frailty | From 3-4 months post enrollment (before surgery) (T2) to 4-7 months post enrollment (90 days post surgery) (T3)
  Frailty will be assessed using the Cancer and Aging Resilience Geriatric Assessment.
Frailty | From enrollment (T1) to 4-7 months post enrollment (90 days post surgery) (T3
  Frailty will be assessed using the Cancer and Aging Resilience Geriatric Assessment.
Body composition - fat free mass | From enrollment (T1) to 3-4 months post enrollment (before surgery) (T2)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating the skeletal muscle index and fat mass index of deidentified computed tomography scans.
Body composition - fat free mass | From 3-4 months post enrollment (before surgery) (T2) to 4-7 months post enrollment (90 days post surgery) (T3)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating the skeletal muscle index and fat mass index of deidentified computed tomography scans.
Body composition - fat free mass | From enrollment (T1) to 4-7 months post enrollment (90 days post surgery) (T3)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating the skeletal muscle index and fat mass index of deidentified computed tomography scans.
Body composition - fat mass | From enrollment (T1) to 3-4 months post enrollment (before surgery) (T2)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating fat mass index of deidentified computed tomography scans.
Body composition - fat mass | From 3-4 months post enrollment (before surgery) (T2) to 4-7 months post enrollment (90 days post surgery) (T3)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating fat mass index of deidentified computed tomography scans.
Body composition - fat mass | From enrollment (T1) to 4-7 months post enrollment (90 days post surgery) (T3)
  Body composition will be measured using a validated, supervised machine learning body composition segmentation algorithm evaluating fat mass index of deidentified computed tomography scans.
Patient-reported health-related quality of life | At enrollment, 3-4 months from enrollment (before surgery), 4-7 months from enrollment (90 days post surgery)
  Patient reported health-related quality of life will be assessed by a change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ)-C30. All of the subscales and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale and global health status scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
Patient-reported health-related quality of life - bladder cancer specific | From enrollment (T1) to 3-4 months post enrollment (before surgery) (T2)
  Bladder cancer-specific patient-reported health-related quality of life will be assessed by a change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-Bladder Cancer Muscle-Invasive 30). All subscale and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale and global health status scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
Patient-reported health-related quality of life - bladder cancer specific | From 3-4 months post enrollment (before surgery) (T2) to 4-7 months post enrollment (90 days post surgery) (T3)
  Bladder cancer-specific patient-reported health-related quality of life will be assessed by a change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-Bladder Cancer Muscle-Invasive 30). All subscale and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale and global health status scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
Patient-reported health-related quality of life - bladder cancer specific | From enrollment (T1) to 4-7 months post enrollment (90 days post surgery) (T3)
  Bladder cancer-specific patient-reported health-related quality of life will be assessed by a change in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC-QLQ-Bladder Cancer Muscle-Invasive 30). All subscale and single-item measures range in score from 0 to 100 and a high scale score represents a higher response level (ranging from 0 = low to 100 = high/healthy level of function; from 0 = low to 100 = high quality-of-life; from 0 = low to 100 = high level of symptomatology/problems). Subscale and global health status scores are each calculated by transforming individual item scores into a 0 to 1 scale, taking the mean, and multiplying by 100.
NAC-associated adverse events | From enrollment (T1) to 3-4 months post enrollment (before surgery) (T2)
  Will be recorded as both physician-reported adverse events utilizing Common Terminology Criteria for Adverse Events (CTCAE), version (v.) 5.0 and using the patient-reported CTCAE and will be described via qualitative report
(P)REHAB-associated adverse events | At enrollment (T1), 3-4 months from enrollment (before surgery) (T2), 4-7 months from enrollment (90 days post surgery) (T3)
  Will be assessed by comparing physician-reported CTCAE v. 5.0 adverse events (e.g. falls, pain score as measured using a visual analog scale 0-10, and fatigue), compared between the (P)REHAB and standard of care arms.
Number of participants with post-surgical complications within 90 days graded using the Clavien grading scale | Within 90 days of surgery
  Graded using the Clavien grading scale and reported qualitatively. The Clavien-Dindo Classification is a grading system used throughout surgery for classifying adverse events (complications) that occur as a result of surgical procedures. The system consists of five (I, II, III, IV and V) or seven (I, II, IIIa, IIIb, IVa, IVb and V) grades of severity, with Grade I being low and Grade V being death.
Surgical outcomes - length of stay | Through study completion, on average 7 months
  Surgical outcomes include length of stay following surgery. Surgical outcomes will be reported via qualitative report.
Surgical outcomes - post discharge disposition | Through study completion, on average 7 months
  Surgical outcomes include discharge disposition (e.g. discharge to home vs. short term nursing facility versus rehabilitation unit). For patients not discharged to home, will evaluate length of time in a skilled nursing facility or rehabilitation unit as necessary. Surgical outcomes will be reported via qualitative report
Average daily step count | Through study completion, on average 7 months
  Number of steps per day as measured by the FitBit wearable will be reported.
Average daily sedentary time | Through study completion, on average 7 months
  Average daily sedentary time as measured by the FitBit wearable will be reported.
Provider perceived usability | Up to 1 year
  Assessed using the System Usability Scale (SUS) score 0-100 with 100 being high usability, User Burden Scale (UBS) score 20-100 with 100 being high burden, and/or Intervention Usability Scale (IUS) score 0-100 with 100 being high usability.
Provider perceived utility | Up to 1 year
  Assessed using the System Usability Scale (SUS) score 0-100 with 100 being high usability, User Burden Scale (UBS) score 20-100 with 100 being high burden, and/or Intervention Usability Scale (IUS) score 0-100 with 100 being high usability.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Psutka, Principal Investigator — Fred Hutch/University of Washington Cancer Consortium
Locations (1):
- Fred Hutch/University of Washington Cancer Consortium, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhu A, Sher J, Li R, Ioseliani O, Cantor L, Brewer EG, Landis K, Bridges D, Munson SA, Hunter H, Lin C, Psutka SP. What motivates bladder cancer patients to be active? A qualitative study assessing attitudes towards physical activity and digital health technologies. Urol Oncol. 2025 Sep;43(9):522.e1-522.e8. doi: 10.1016/j.urolonc.2025.05.002. Epub 2025 May 28. PMID 40441948